CLINICAL TRIAL: NCT04712006
Title: Phase 1, Open-label, Single Dose Study to Investigate the Pharmacokinetics, Safety, and Tolerability of JNJ-64304500 Following Subcutaneous Injection in Healthy Chinese Adult Participants
Brief Title: A Study of JNJ-64304500 Following Subcutaneous Injection in Healthy Chinese Adult Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108840; 64304500CRD1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: JNJ-64304500 (Experimental): Participants will receive single subcutaneous (SC) Dose 1 of JNJ-64304500 on Day 1.
  Interventions: Drug: JNJ-64304500
- Cohort 2: JNJ-64304500 (Experimental): Participants will receive single SC Dose 2 of JNJ-64304500 on Day 1.
  Interventions: Drug: JNJ-64304500

INTERVENTIONS:
Drug: JNJ-64304500 — Participants will be administered with JNJ-64304500 SC (Dose 1 or 2) injection on Day 1.

SUMMARY:
The purpose of this study is to assess the pharmacokinetic following single subcutaneous administration of Dose 1 or Dose 2 of JNJ-64304500 in healthy Chinese adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese participants whose parents and maternal and paternal grandparents are of Chinese ethnicity
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and until Day 113
* A male participant must agree not to donate sperm for the purpose of reproduction and must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and until Day 113
* A woman must have a negative highly sensitive serum beta-human chorionic gonadotropin (hCG) at screening and a negative urine pregnancy test on Day -1 and while enrolled in this study
* Nonsmoker or agree to smoke no more than 10 cigarettes or equivalent of e-cigarettes, or 2 cigars, or 2 pipes of tobacco per day throughout the study, if the inpatient unit allows. However, if smoking is not allowed in the inpatient unit, smokers will not be allowed to smoke while inpatient and cannot use nicotine replacement products during the inpatient period

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should be exclude the participant, including (but not limited to) liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Had major illness or surgery, (example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from illness or surgery, or has surgery planned during the time the participant is expected to participate in the study or until Day 113
* Plans to undergo non-major elective surgery within 4 weeks prior to study intervention administration through the end of the study
* Known or suspected allergies, hypersensitivity or intolerance to JNJ-64304500 or any biologic medication, or known allergies or clinically significant reactions to murine, chimeric, or human proteins, mAbs or antibody fragments, or to any components of the formulation of JNJ-64304500 and its excipients used in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-30 (Estimated); Primary Completion 2021-08-27 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Serum Concentration of JNJ-64304500 | Up to Day 113
  Serum samples will be analyzed to determine concentrations of JNJ-64304500 using a validated, specific and sensitive immunoassay method.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 113
  An AE is any untoward medical occurrence in a clinical study participant administered an investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.
Number of Participants with Antibodies to JNJ-64304500 | Up to Day 113
  Number of participants with antibodies to JNJ-64304500 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency